CLINICAL TRIAL: NCT05240638
Title: Feasibility of Transcatheter Cannulation and Drainage of the Thoracic Duct in Patients With Congestive Heart Failure
Brief Title: Lymph Drainage in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00107814
Record Dates: First submitted 2022-01-10; First posted 2022-02-15 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
Keywords: heart catheterization; heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TD Drainage (Experimental): Short term TD drainage
  Interventions: Device: TD Drainage

INTERVENTIONS:
Device: TD Drainage — Image-guided percutaneous cannulation of the TD and drainage with an endovascular catheter (microcatheter)

SUMMARY:
This study aims to test the safety and efficacy of lymph fluid drainage on heart congestion and shortness of breath symptoms among patients participants with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Subjects with informed consent to participate
* NYHA III- IV patients
* Patients with heart failure volume overload
* Planned for elective right heart catheterization

Exclusion Criteria:

* Active coronary syndrome (type I myocardial infarction)
* Local infection or ongoing systemic infection(s)
* Thrombotic coagulation disorder
* On continuous blood thinners that cannot be discontinued or held
* Allergy or contraindications to the use of iodine-based contrast agents
* Subjects deemed to be high risk for performing a cardiac catheterization by study investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Technical success for access | At the time of the procedure
  Number of patients where TD was accessed successfully with an endovascular catheter under fluoroscopic or ultrasound guidance
Safety defined as the absence of serious adverse events | Up to 24 hours post-procedure
  Safety as measured by number of serious adverse events
Technical success for drainage | At the time of the procedure
  Number of patients where any amount of lymph was drained successfully from the TD with an endovascular catheter

SECONDARY OUTCOMES:
Total fluid output (measured in mL) as measured by fluid collection | Up to 24 hours post-procedure
  Total fluid output (measured in mL) as measured by fluid collection
Change in body weight | Pre-procedure, Post-procedure (up to 4 hours)
  Change in body weight
Change in blood N-terminal Pro-BNP as measured by lab test | Baseline, 12 hours, 24 hours post initiation of drainage
  Change in blood N-terminal Pro-BNP as measured by lab test
Number of HF-related hospitalizations as measured by medical record review | 30 days post-discharge
  Number of HF-related hospitalizations as measured by medical record review

CONTACTS AND LOCATIONS:
Overall Officials: Marat Fudim, MD, Principal Investigator — Duke University
Locations (1):
- Marat Fudim, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No